CLINICAL TRIAL: NCT02390297
Title: Long Term Follow-up for the Detection of Delayed Adverse Events in Recipients of CD4+ T Lymphocytes and/or CD34+ Hematopoietic Stem/Progenitor Cells Transduced With LVsh5/C46, a Dual Anti-HIV Gene Transfer Construct
Brief Title: Long Term Follow up for the Detection of Delayed Adverse Events in Cal-1 Recipients
Status: Active, not recruiting | Type: Observational
Sponsor: Calimmune, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAL-INT-00
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: HIV-1 Infection; Receipt of Cal-1 Modified Hematopoietic Cellular Products
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cryopreserved white blood cells and DNA and RNA extracted from peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single: Collection of blood samples for general health (complete blood count) and Cal-1 specific analyses
  Interventions: Genetic: Blood tests

INTERVENTIONS:
Genetic: Blood tests — Collection of blood samples for general health (complete blood count) and Cal-1 specific analyses

SUMMARY:
Long term safety follow-up of Cal-1 recipients

DETAILED DESCRIPTION:
Long Term Follow-up for the Detection of Delayed Adverse Events in Recipients of CD4+ T Lymphocytes and/or CD34+ Hematopoietic Stem/Progenitor Cells Transduced with LVsh5/C46 (Cal-1), a Dual Anti-HIV Gene Transfer Construct

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Previous treatment with the Cal-1 modified hematopoietic cellular products

Exclusion Criteria:

* Inability to understand and provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligibility for this protocol is dependent on prior exposure to a Cal-1 modified hematopoietic cellular product. The study population will thus consist of individuals with HIV-1 infection, who have met criteria for participation in a Cal-1 phase I/II clinical trial and received a dose of Cal-1 modified hematopoietic cells as part of a previous study
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Detection of delayed clinical or molecular adverse events related to Cal-1, or the associated delivery procedures | 15 years

SECONDARY OUTCOMES:
Assessment of the long term survival and activity of Cal-1 modified hematopoietic cells through evaluation of Cal-1 marking and expression in peripheral blood | 15 yars

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Landovitz, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA CARE Center, Los Angeles, California
  - Quest Clinical Research, San Francisco, California